CLINICAL TRIAL: NCT05125341
Title: Natural History Study of Adult Patients With Paroxysmal Nocturnal Hemoglobinuria of High-risk Hemolysis in China
Status: Completed | Type: Observational
Sponsor: CARE Pharma Shanghai Ltd. (Industry)
Responsible Party: Sponsor
Organization: CANbridge Life Sciences Ltd. (Industry)
Other Study IDs: CAN106-01001
Record Dates: First submitted 2021-11-08; First posted 2021-11-18 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2021-11

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria, Natural History Study
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a single-center observational study conducted in adult patients with paroxysmal nocturnal hemoglobinuria of high-risk hemolysis.

This observational study consists of two parts, one part is retrospective study which aims to collect medical chart data to calculate the mean change or mean incidence rates of LDH, hemoglobin, PNH-related symptoms and PNH-related events over 6 months.

The other part is cross-sectional study to detect the total C5 level in PUMCH at the latest follow-up visit in eligible PNH patients with high-risk hemolysis, to show the difference between eligible PNH patients and healthy people and to explore the related clinical factor influencing high-level total C5 using logistic regression model.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for paroxysmal nocturnal hemoglobinuria;
2. Age ≥ 18 years old;
3. PNH clone size of granulocytes or monocytes (CD59 or Flaer) ≥ 10%;
4. LDH≥1.5 ULN;
5. Accompanied by at least one PNH-related symptoms: fatigue, hemoglobinuria, abdominal pain, dyspnea, anemia symptoms, major adverse vascular events (including thrombosis), dysphagia, erectile dysfunction;
6. Transfusion-dependent PNH patients;
7. There are at least 6 months consecutive data of diagnosis and treatment after the data collection time point;
8. Patients agreed to participate in the study by signing informed consent or giving oral informed consent.

Exclusion Criteria:

1. Patients are under the treatment of the C1/C3/C5 complement inhibitors currently or in the past;
2. Patients have received bone marrow transplantation;
3. platelet count <30*10 9/L or absolute neutrophil count <0.5*10 9/L;
4. Patients have clinically significant heart, liver, or lung diseases, or have related medical history.
5. Patients have comorbidities of rheumatoid disease, HIV infection, active HBV infection, HCV infection and other diseases that affect the body's immune function;
6. Severe missing data in the records of diagnosis and treatment after the data collection time point;
7. Other patients who are not suitable to participate in the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with paroxysmal nocturnal hemoglobinuria of high-risk hemolysis in China
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
the mean change of LDH | 6 months
  the mean change of LDH over 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bing Han, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China